CLINICAL TRIAL: NCT05619952
Title: Acute Effects of White Button and Shiitake Mushroom Powder Supplementation on Postprandial Lipemia and Glycemia Following a High-Fat Meal
Brief Title: Postprandial Lipemia and Glycemia Following a High-Fat Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Lillian A. Talal, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 030-614292
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Hypercholesterolemia; Postprandial Hyperglycemia; Lipid Disorder
Keywords: mushroom; lipid metabolism; postprandial lipemia; postprandial glycemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperglycemia; Lipid Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind, randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- White Button Mushroom (Experimental): 368.5 grams of irradiated ground beef patty (80/20 lean mass to fat ratio) + 14 grams white button mushroom powder, and a Wegmans Food Market Brand Big Hawaiian bun
  Interventions: Dietary Supplement: Mushroom Powder
- Shiitake Mushroom (Experimental): 368.5 grams of irradiated ground beef patty (80/20 lean mass to fat ratio) + 14 grams Shiitake mushroom powder, and a Wegmans Food Market Brand Big Hawaiian bun
  Interventions: Dietary Supplement: Mushroom Powder
- Control (No Intervention): 368.5 grams of irradiated ground beef patty (80/20 lean mass to fat ratio) and a Wegmans Food Market Brand Big Hawaiian bun.

INTERVENTIONS:
Dietary Supplement: Mushroom Powder — Ground shiitake mushrooms or ground white button mushrooms
  Arms: Shiitake Mushroom; White Button Mushroom

SUMMARY:
The goal of this clinical trial is to determine the acute effects on postprandial lipemia and glycemia by supplementing a high-fat meal with either white button (WB) or shiitake (SH) mushroom powder in relatively healthy adults, aged 18 to 35.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* non-diabetic
* normal to mildly hypercholesterolemic (Total Cholesterol 200-239 mg/dL and LDL-C 130-159 mg/dL)
* have BMI <30 or BF% (men <25%, women <32%)
* no known disease of the liver or gallbladder
* no documented problems with fat metabolism
* normal lipemic response to a lipid challenge
* No known mushroom allergy

Exclusion Criteria:

* diabetic
* pregnant
* BMI >30
* liver disease
* gallbladder disease
* mushroom allergy
* lipid disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12-29 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Postprandial Lipemia | Baseline, up to 6 hours postprandial
  Total cholesterol, LDL, HDL, triglycerides
Postprandial Glycemia | Baseline, up to 6 hours postprandial
  blood glucose

REFERENCES:
- [Result] Lillian A. Talal, Huipei Wang, Brian T. Wil-liams, Matthew J. Morris, Peter J. Horvath (2023) Acute Effects of White Button and Shiitake Mushroom Powder Supplementa-tion on Postprandial Lipemia and Glycemia Following a High-Fat Meal . International Journal of Nutrition - 7(2):42-56.
- See also: Related Info — https://doi.org/10.14302/issn.2379-7835.ijn-23-4430